CLINICAL TRIAL: NCT06083168
Title: Cardiovascular Disease in Patients With Chronic Kidney Disease: Polish Kidney- Heart Project
Status: Recruiting | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: University of Warmia and Mazury in Olsztyn (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: Polish Kidney-Heart Project
Record Dates: First submitted 2023-09-08; First posted 2023-10-13 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Disease; Cardiovascular Diseases
Keywords: chronic kidney disease; cardiovascular disease; artificial inteligence; predictors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational longitudinal study which will collect routine demographic, laboratory and clinical parameters of patients with chronic kidney disease (CKD) in the Silesian and Warmia and Mazury Regions (Poland) aimed at predicting incident cardiovascular disease and cardiovascular and renal events using machine learning and artificial intelligence approaches. There will be a subgroup analysis of patients with diabetes and CKD.

DETAILED DESCRIPTION:
This is a prospective, observational study seeking to collate demographic, laboratory, and clinical data from patients with CKD hospitalized at two academic centres: the Department of Internal Medicine, Diabetology and Nephrology in Zabrze, Silesia, and the Clinic of Nephrology, Hypertension and Internal Medicine in Olsztyn, Warmia and Mazury.

Patients will receive telephone check-ups annually post-discharge and will be proposed to attend on-site follow-up health checks. Patients will be followed up annually for 10 years or until death if occurs earlier, in order to collect information related to new onset cardiovascular events and progression to macroalbuminuria and/or doubling of serum creatinine with decrease of eGFR to less than 45 ml/min./1.73m2 (compared to baseline) or the onset of end stage renal disease (ESRD) or renal death. ESRD is defined as initiation of maintenance dialysis or kidney transplantation. All procedures, except eye fundus imaging for hospitalized patients align with standard nephrology ward care that patients agree for upon hospitalization.

The Medical University of Silesia and the University of Warmia and Mazury, Collegium Medicum obtained study approvals from the respective independent university- or chamber of physicians-based bioethics committees for performing fundus imaging during hospital stay and annual telephone contacts as well as on- site health checks for the longitudinal patient follow-up observation.

With patient consent, annual on-site visits will entail blood and urine assessments, ECG, retinal imaging via the fundus camera, and examinations for peripheral and cardiac autonomic neuropathy among those with diabetes. Biochemical analyses will focus on assessing serum creatinine, lipid profile, HbA1c for diabetic patients, and the urine albumin-creatinine ratio (UACR).

With a decade-long prospective follow-up focused on documenting new cardiovascular and renal events, the primary objective is to identify patients with CKD at the highest risk of cardiovascular disease and CKD progression. This goal will be achieved by implementing machine learning techniques to analyze clinical parameters that are easy to obtain in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* CKD defined as estimated glomerular filtration rate (eGFR) < 60ml/min/1.73 m2 and/or urine albumin creatinine ratio ( UACR) > 30 mg/g lasting at least 3 months
* CKD regardless of eGFR/albuminuria when documented otherwise (by means of imaging, renal biopsy result, genetic background, etc)

Exclusion Criteria:

* Death during hospital stay
* Terminal stage of cancer
* Lack of an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in nephrology departments in Zabrze and Olsztyn.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2033-11-30 (Estimated); Study Completion 2036-01-31 (Estimated)

PRIMARY OUTCOMES:
Incident Coronary Artery Disease | Annually, 10 years from enrollment
  New occurrence of coronary artery disease as diagnosed by standard medical procedures.
Myocardial Infarction | Annually, 10 years from enrollment
  New occurrence of myocardial infarction as confirmed by electrocardiogram and/or biomarkers.
New onset heart failure or exacerbation of heart failure | Annually, 10 years from enrollment
  New-Onset Heart Failure: Diagnosis based on the ESC guidelines, which include symptoms such as breathlessness, ankle swelling, and fatigue; objective evidence of cardiac dysfunction or structural abnormality in echocardiography; and response to treatment directed towards heart failure.
  Hospitalization for decompensated heart failure: Requires unscheduled admission to a healthcare facility with heart failure as the primary reason for admission.
Stroke or Transient Ischemic Attack | Annually, 10 years from enrollment
  New occurrence of stroke as confirmed by neuroimaging or transient ischemic attack ascertained by typical symptoms.
Peripheral Vascular Disease Peripheral Vascular Disease Peripheral Vascular Disease Peripheral Vascular Disease Peripheral Vascular Disease | Annually, 10 years from enrollment
  New diagnosis of peripheral vascular disease confirmed by imaging studies.
Atrial Fibrillation | Annually, 10 years from enrollment
  Incident atrial fibrillation confirmed by electrocardiogram.
Death Due to Cardiovascular Cause | Annually, 10 years from enrollment
  Death where the primary cause is attributed to cardiovascular disease.
Progression of Chronic Kidney Disease | Annually, 10 years from enrollment
  Progression to macroalbuminuria or doubling of serum creatinine with a decrease of eGFR to less than 45 ml/min/1.73m^2 compared to baseline.
End-Stage Renal Disease or Renal Death | Annually, 10 years from enrollment
  Onset of end-stage renal disease requiring initiation of maintenance dialysis or kidney transplantation, or death due to renal causes.

SECONDARY OUTCOMES:
Machine-learning predictors of outcomes, including ECG predictors and retinal imaging predictors. | 10 years from enrollment
  Using new statistical methods in predicting outcomes
Cluster analyses. | 10 years from enrollment
  Use of statistical cluster analysis to identify patterns within primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Nabrdalik, assoc. Prof, Principal Investigator — Medical University of Silesia; Tomasz Stompór, Prof., Principal Investigator — The University of Warmia and Mazury in Olsztyn; Gregory YH Lip, Prof., Study Chair — University of Liverpool; Janusz Gumprecht, Prof., Study Chair — Medical University of Silesia
Locations (2):
- Poland (2):
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. prof. Stanisława Szyszko Śląskiego Uniwersytetu Medycznego w Katowicach, Zabrze

IPD SHARING:
Plan to Share IPD: No